CLINICAL TRIAL: NCT01476670
Title: Cerebral Autoregulation and Carbon Dioxide Reactivity in Patients With Posterior Fossa Tumor
Brief Title: Cerebral Blood Circulation in Patients With Posterior Fossa Brain Tumor
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hemanshu Prabhakar, Dr., All India Institute of Medical Sciences
Other Study IDs: CA-CO2-TCD; Posterior fossa tumor - TCD (Other: AIIMS)
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Last update posted 2011-11-22 (Estimated); Status verified 2011-11

CONDITIONS: Brain Tumor
Keywords: Posterior fossa brain tumor; Cerebral blood flow; Cerebral autoregulation; Carbon dioxide reactivity; Transcranial Doppler
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Posterior fossa tumor: Patients with posterior fossa tumor scheduled for elective surgery will be enrolled in the study.
  Interventions: Other: Monitoring

INTERVENTIONS:
Other: Monitoring — Transcranial Doppler will be used to assess the cerebral autoregulation and carbon dioxide reactivity of patients with posterior fossa tumor

SUMMARY:
The normal cerebral blood flow is guided by factors such as cerebral autoregulation (CA) and carbon dioxide reactivity (CO2R). Authors have demonstrated that CA and CO2R may be impaired in presence of intracranial tumors.Most studies pertaining to assessment of CA and CO2R in patients with brain tumors is limited to supratentorial tumors. Due to their anatomic location, posterior fossa tumors result in obstruction of ventricular outflow, produce hydrocephalus and features of raise intracranial pressure (ICP). It is possible that lesions in the posterior fossa may affect CA and CO2R. It should also be noted that posterior fossa surgeries are carried out in positions such as prone, lateral and sitting. Altered surgical positions themselves affect systemic hemodynamics which may influence cerebral blood flow; with presence of anesthetics further compromising the blood flow to the brain. Understanding the homeostatic mechanisms of CA and CO2R may help in deciding proper positioning of patients and maintenance of intraoperative hemodynamic.

The aim of this observational study was to evaluate CA and CO2R in patients with posterior fossa tumor prior to surgical decompression of the lesion.

ELIGIBILITY:
Inclusion Criteria:

* All patients with posterior fossa tumor
* Scheduled for elective surgery
* History of recent ventriculoperitoneal shunt (within 24 hours)

Exclusion Criteria:

* previous craniotomy
* patients on ventilatory support
* history of cerebrovascular accident
* syncope or carotid artery disease
* anemia
* polycythemia
* patients on vasoactive medications
* those suffering from medical conditions such as diabetes mellitus and hypertension.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Due to their anatomic location, posterior fossa tumors result in obstruction of ventricular outflow, produce hydrocephalus and features of raise intracranial pressure (ICP). It is possible that lesions in the posterior fossa may affect Cerebral Autoregulation and Carbon dioxide reactivity. It should also be noted that posterior fossa surgeries are carried out in positions such as prone, lateral and sitting. Altered surgical positions themselves affect systemic hemodynamics which may influence cerebral blood flow; with presence of anesthetics further compromising the blood flow to the brain. Understanding the homeostatic mechanisms of CA and CO2R may help in deciding proper positioning of patients and maintenance of intraoperative hemodynamic.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-07

CONTACTS AND LOCATIONS:
Overall Officials: Hemanshu Prabhakar, MD, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi, India